CLINICAL TRIAL: NCT05994768
Title: Comparison of the Performance of 18F-FDG PET/CT With That of Labeled Leukocyte Scintigraphy in the Follow-up of Malignant Otitis Externa.
Brief Title: 18F-FDG Tomography and Labeled Leukocyte Scintigraphy
Acronym: OEN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2023PI003
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Malignant Otitis Externa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 18F-FDG PET/CT — Patients who underwent an 18F-FDG PET/CT examination and a labeled leukocyte scintigraphy before and after antibiotic therapy in the case of management of an EO.
  Other Names: scintigraphy with labeled leukocytes

SUMMARY:
The study will aim to show that there is a superiority of 18F-FDG PET/CT compared to labeled leukocyte scintigraphy in patients with a malignant otitis externa.

DETAILED DESCRIPTION:
The management of malignant otitis externa (MEO) is a major issue in patients who are often polypathological and fragile. Appropriate antibiotic therapy must be started quickly after the diagnosis is made and followed for a period of at least 6 weeks. Imaging plays a major role in assessing the extent of the infection and especially healing, after 6 weeks of antibiotic therapy. The persistence of an infection at the end of the treatment, observed in imaging, will allow a change of antibiotic line. This study consists in studying in a population affected by an OEM, the performance of PET/CT with 18F-FDG compared to scintigraphy with labeled leukocytes. The usefulness of the latter in the follow-up of the pathology after antibiotic therapy has already been proven in the literature. The study will aim to show that there is a superiority of 18F-FDG PET/CT compared to labeled leukocyte scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant otitis externa who received a 18F-FDG positron emission tomography and a labelled leukocyte scintigraphy

Exclusion Criteria:

* patients who refuse to have their imaging data used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent an 18F-FDG positron emission tomography examination and a labeled leukocyte scintigraphy before and after antibiotic therapy in the case of management of an malignant otitis externa.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
18F-FDG positron emission tomography | one day
  measurement of standard uptake value
Labeled leukocyte scintigraphy | one day
  measurement of standard uptake value

CONTACTS AND LOCATIONS:
Locations (1):
- Verger Antoine, Vandœuvre-lès-Nancy, France